CLINICAL TRIAL: NCT00916110
Title: Ascending Single Dose Study Of The Safety, Tolerability, PK And PD Of ATN-103 Administered SC Or IV To Healthy Japanese Male Subjects
Brief Title: Study Of Single Dose Of ATN-103 Administered To Healthy Japanese Male Subjects
Acronym: ATN-103
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3242K1-1001; B2271002
Record Dates: First submitted 2009-05-28; First posted 2009-06-09 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: healthy subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- 1.5mgSC (Experimental): ATN-103
  Interventions: Drug: ATN-103
- 4mgSC (Experimental): ATN-103
  Interventions: Drug: ATN-103
- 10mgSC (Experimental): ATN-103
  Interventions: Drug: ATN-103
- 25mgSC (Experimental): ATN-103
  Interventions: Drug: ATN-103
- 25mgIV (Experimental): ATN-103
  Interventions: Drug: ATN-103
- 50mgSC (Experimental): ATN-103
  Interventions: Drug: ATN-103
- 100mgSC (Experimental): ATN-103
  Interventions: Drug: ATN-103
- 200mgSC (Experimental): ATN-103
  Interventions: Drug: ATN-103
- 200mgIV (Experimental): ATN-103
  Interventions: Drug: ATN-103

INTERVENTIONS:
Drug: ATN-103 — 1.5 mg solution, single subcutaneous injection
  Arms: 1.5mgSC
Drug: ATN-103 — 4 mg solution, single subcutaneous injection
  Arms: 4mgSC
Drug: ATN-103 — 10 mg solution, single subcutaneous injection
  Arms: 10mgSC
Drug: ATN-103 — 25 mg solution, single subcutaneous injection
  Arms: 25mgSC
Drug: ATN-103 — 25 mg solution, single intravenous injection
  Arms: 25mgIV
Drug: ATN-103 — 50 mg solution, single subcutaneous injection
  Arms: 50mgSC
Drug: ATN-103 — 100 mg solution, single subcutaneous injection
  Arms: 100mgSC
Drug: ATN-103 — 200 mg solution, single subcutaneous injection
  Arms: 200mgSC
Drug: ATN-103 — 200 mg solution, single intravenous injection
  Arms: 200mgIV

SUMMARY:
To assess the safety and tolerability of ascending single SC and IV doses of ATN-103 in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male subjects aged 20 to 45 with health determined by the study investigator.
* BMI in the range of 17.6 to 26.4.
* Nonsmoker or male who smokes fewer than 10 cigarettes per day.

Exclusion Criteria:

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Acute disease state (eg, nausea, vomiting, infection, fever, or diarrhea) within 7 days before study day 1.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability are evaluated from the reported AEs, vital sign, laboratory test, etc. | 24weeks

SECONDARY OUTCOMES:
Antibody in blood and drug concentration in blood and urine are evaluated. | 24weeks

CONTACTS AND LOCATIONS:
Overall Officials: Josefin-Beate Holz, MD, Study Director — Ablynx NV
Locations (1):
- Investigational Site, Toshima City, Tokyo, Japan